CLINICAL TRIAL: NCT01566188
Title: Cardiovascular Impact of Omega-3 Dietary Supplement From Vegetal Origin in Hypertension Associated With Metabolic Syndrome
Brief Title: Vascular Impact of Omega-3 in Metabolic Syndrome
Acronym: CARDIOMEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 2010/010 HP
Record Dates: First submitted 2011-12-08; First posted 2012-03-29 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Essential Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Essential Hypertension; Metabolic Syndrome | interventions — Cyclodextrins; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omega-3 from vegetal origin (Experimental)
  Interventions: Dietary Supplement: omega-3 from vegetal origin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 from vegetal origin — 6 months of supplementation with omega-3 from vegetal origin
  Other Names: Cyclodextrin/Camelin oil
  Arms: omega-3 from vegetal origin
Dietary Supplement: Placebo — 6 months of supplementation with placebo
  Other Names: Cyclodextrin/Starch
  Arms: Placebo

SUMMARY:
The overall aims of the present project are to investigate the impact of a nutritional approach based on omega-3 from vegetal origin on vascular function in hypertension associated with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with treated essential hypertension (blood pressure values<140/90 mmHg under antihypertensive treatment).
* Presence of at least two of the following criteria of the metabolic syndrome: abdominal girth >102 cm in men or >88 cm in women, HDL-C<0.4 g/L in men or <0.5 g/L in women, fasting triglyceride >1.5 g/L (or specific treatment for these lipid abnormalities), fasting glucose >1.10 g/L.

Exclusion Criteria:

* Secondary hypertension, myocardial infarction, coronary artery disease, cerebrovascular disease, stroke or transient ischemia, cardiac failure, diabetes (or fasting glucose>1.26 g/L) or renal failure (MDRD < 50 ml/min)
* Severe hypercholesterolemia (total cholesterol > 2.5 g/l), alcohol or drug abuse, toxicomania, or clinically significant abnormalities in other current biological parameters.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilatation | 6 months after omega-3 supplementation

SECONDARY OUTCOMES:
Aortic stiffness | 6 months after omega-3 supplementation
  carotid-to-femoral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Robinson Joannides, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Mahes Hospital, Fleury-Mérogis
  - George Pompidou European Hospital, Paris
  - Rouen University Hospital, Rouen
  - Rangueil University Hospital, Toulouse